CLINICAL TRIAL: NCT01900665
Title: Effect of Passive Immunization on the Progression of Mild Alzheimer's Disease: Solanezumab (LY2062430) Versus Placebo
Brief Title: Progress of Mild Alzheimer's Disease in Participants on Solanezumab Versus Placebo
Acronym: EXPEDITION 3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Solanezumab did not meet the study's primary endpoint.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15136; H8A-MC-LZAX (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — solanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solanezumab (Experimental): Solanezumab 400 milligrams (mg) every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who complete the full 80 weeks of treatment/assessment and decide to continue will take this regimen for up to an additional 208 weeks.
  Interventions: Drug: Solanezumab
- Placebo (Placebo Comparator): Placebo every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who complete the full 80 weeks of treatment/assessment and decide to continue will switch to solanezumab 400 mg every 4 weeks for up to an additional 208 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solanezumab — Administered Intravenously (IV)
  Other Names: LY2062430; A Beta Antibody
  Arms: Solanezumab
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
To test the idea that solanezumab will slow the cognitive decline of Alzheimer's Disease (AD) as compared with placebo in participants with mild AD.

ELIGIBILITY:
Inclusion Criteria:

* Meets National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable AD
* Has a Modified Hachinski Ischemia Scale score of less than or equal to 4
* Has a Mini-Mental State Examination (MMSE) score of 20 through 26 at Screening visit
* Has a Geriatric Depression Scale score of less than or equal to 6 (on the staff-administered short form)
* Has had a magnetic resonance imaging (MRI) or computerized tomography (CT) scan performed within the past 2 years that has confirmed no findings inconsistent with a diagnosis of AD
* Has a florbetapir positron emission tomography (PET) scan or cerebrospinal fluid (CSF) result consistent with the presence of amyloid pathology at screening

Exclusion Criteria:

* Does not have a reliable caregiver who is in frequent contact with the participant (defined as at least 10 hours per week), will accompany the participant to the office and/or be available by telephone at designated times, and will monitor administration of prescribed medications
* Meets National Institute of Neurological Disorders and Stroke/Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS/AIREN) criteria for vascular dementia
* Has current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study; or has a life expectancy of <2 years
* Has had a history within the last 5 years of a serious infectious disease affecting the brain or head trauma resulting in protracted loss of consciousness
* Has a history within the last 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate-specific antigen posttreatment
* Has a known history of human immunodeficiency virus (HIV), clinically significant multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions
* Has received acetylcholinesterase inhibitor (AChEIs), memantine and/or other AD therapy for less than 4 months or has less than 2 months of stable therapy on these treatments
* Has received medications that affect the central nervous system (CNS), except treatments for AD, for less than 4 weeks
* Has a history of chronic alcohol or drug abuse/dependence within the past 5 years
* Has a Visit 1 MRI with results showing >4 Amyloid-related Imaging Abnormality (ARIA), -hemorrhage /hemosiderin deposition (ARIA-H) or presence of ARIA-E (edema/effusions)

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2129 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (198):
- United States (120):
  - Xenoscience, Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - ANI Arizona Neurological Institute Research, PC, Sun City, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Arizona Health Sciences Center, Tucson, Arizona
  - American Neuropsychiatric Research Institute, Inc, Carson, California
  - Neurology Center of North Orange County, Fullerton, California
  - Institute for Memory Impairment & Neurological Disorders, Irvine, California
  - University of California - San Diego, La Jolla, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Torrance Clinical Research, Lomita, California
  - Collaborative Neuroscience Network - CNS, Long Beach, California
  - Apostle Clinical Trials, Inc, Long Beach, California
  - Univ of Southern California Medical Center, Los Angeles, California
  - University of California Los Angeles School of Medicine, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Anderson Clinical Research, Redlands, California
  - University of California, Davis - Health Systems, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Pacific Research Network Inc, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Apex Research Institute, Santa Ana, California
  - St. Joseph Health, Santa Rosa, California
  - California Neuroscience Research, Sherman Oaks, California
  - Radiant Research, Denver, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Norwalk, Connecticut
  - Christiana Care Research Institute, Newark, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders, Boca Raton, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Cohen Medical Associates P.A., Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Galiz Research, Hialeah, Florida
  - Infinity Clinical Research . LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mayo Clinic of Jacksonville, Jacksonville, Florida
  - Miami Jewish Home and Hospital for the Aged, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, Orlando, Florida
  - Neurology Clinical Research, Inc, Sunrise, Florida
  - Axiom Research, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - CTT Consultants, Prairie Village, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Baptist Physician's Lexington, Lexington, Kentucky
  - Private Office: J. Gary Booker, Shreveport, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Maine Neurology, Scarborough, Maine
  - PharmaSite Research Inc, Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Northern Michigan Neurology, Traverse City, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Univ of Nebraska Med Center, Omaha, Nebraska
  - Cleveland Clinic of Las Vegas, Las Vegas, Nevada
  - Las Vegas Radiology, Las Vegas, Nevada
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Albuquerque Neurosciences, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Dent Neurological Institute, Amherst, New York
  - SPRI Clinical Trials, LLC., Brooklyn, New York
  - New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Richmond Behavorial Associates, Staten Island, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Behavioral Health Center Research, Charlotte, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Valley Medical Research, Centerville, Ohio
  - Ohio State Univ College Of Medicine, Columbus, Ohio
  - Neurology Specialists Inc., Dayton, Ohio
  - Insight Clinical Trials, Shaker Heights, Ohio
  - Red River Medical Center, LLC, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Summit Research Network Inc, Portland, Oregon
  - Drexel University College of Medicine at EPPI, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Radiant Research, Greer, South Carolina
  - University Psychiatry Associates Avera Health, Sioux Falls, South Dakota
  - Quillen College of Medicine, East TN State University, Johnson City, Tennessee
  - Vanderbilt Univeristy School of Medicine, Nashville, Tennessee
  - Texas Neurology, PA, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Diagnostic Research Group, San Antonio, Texas
  - Radiant Research, Murray, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
  - National Clinical Research - Norfolk Inc, Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Blue Ridge Research Center, Roanoke, Virginia
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington
- Australia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darlinghurst, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Gosford, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caulfield, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fitzroy, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Subiaco, Western Australia
- Canada (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gatineau, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenfield Park, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- France (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reims
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villeurbanne
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Böblingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westerstede
- Italy (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponderano (BI)
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Japan (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barakaldo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guipuzcoa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plasencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt-Girona
- Sweden (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jönköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mölndal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå
- United Kingdom (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath, Avon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Devon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crowborough, East Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scotland, Glasgow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greater London, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salford, Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swindon, Wiltshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Holdridge KC, Yaari R, Hoban DB, Andersen S, Sims JR. Targeting amyloid beta in Alzheimer's disease: Meta-analysis of low-dose solanezumab in Alzheimer's disease with mild dementia studies. Alzheimers Dement. 2023 Oct;19(10):4619-4628. doi: 10.1002/alz.13031. Epub 2023 Mar 22. PMID 36946603
- [Derived] Honig LS, Vellas B, Woodward M, Boada M, Bullock R, Borrie M, Hager K, Andreasen N, Scarpini E, Liu-Seifert H, Case M, Dean RA, Hake A, Sundell K, Poole Hoffmann V, Carlson C, Khanna R, Mintun M, DeMattos R, Selzler KJ, Siemers E. Trial of Solanezumab for Mild Dementia Due to Alzheimer's Disease. N Engl J Med. 2018 Jan 25;378(4):321-330. doi: 10.1056/NEJMoa1705971. PMID 29365294

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded after study enrollment,if PET imaging or CSF results did not show evidence of brain amyloid pathology,a screening MRI with results >4 ARIA-H(amyloid-related imaging abnormality-hemorrhage/hemosiderin deposition) or presence of ARIA-E(amyloid-related imaging abnormality-edema/effusions) and abnormal lab results were found.
Groups:
- Solanezumab: Participants received Solanezumab 400 milligrams (mg)Intravenously (IV) every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who completed the full 80 weeks of treatment/assessment and decide to continue will take this regimen for up to an additional 208 weeks.
- Placebo: Participants received Placebo IV every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who complete the full 80 weeks of treatment/assessment and decide to continue will switch to solanezumab 400 mg every 4 weeks for up to an additional 208 weeks.
Period: Placebo Controlled Period
Arm/Group | Solanezumab | Placebo
Started | 1057 | 1072
Received at Least 1 Dose of Study Drug | 1054 | 1067
Completed | 914 | 908
Not Completed | 143 | 164
Not completed — Death | 9 | 16
Not completed — Adverse Event | 48 | 39
Not completed — Protocol Violation | 1 | 7
Not completed — Withdrawal by Subject | 33 | 45
Not completed — Physician Decision | 11 | 7
Not completed — Lost to Follow-up | 3 | 0
Not completed — Caregiver Decision | 33 | 41
Not completed — Entry Criteria Not Met | 5 | 9
Period: Open Label Period
Arm/Group | Solanezumab | Placebo
Started | 881 (Patients from Placebo Controlled Period were not required to enter into Open Label Period.) | 859 (Patients from Placebo Controlled Period were not required to enter into Open Label Period.)
Completed | 0 | 0
Not Completed | 881 | 859
Not completed — Adverse Event | 16 | 20
Not completed — Death | 5 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Parent/Caregiver Decision | 33 | 34
Not completed — Physician Decision | 4 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor Decision | 802 | 765
Not completed — Withdrawal by Subject | 20 | 28

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Solanezumab: Participants received Solanezumab 400 mg IV every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who completed the full 80 weeks of treatment/assessment and decide to continue will take this regimen for up to an additional 208 weeks.
- Total: Total of all reporting groups
Arm/Group | Solanezumab | Placebo | Total
Number analyzed (Participants) | 1057 | 1072 | 2129
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.69 (7.814) | 73.26 (7.966) | 72.98 (7.894)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 600 | 631 | 1231
  Male | 457 | 441 | 898
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants who had baseline ethnicity data.
  Participants
    number analyzed (Participants) | 970 | 986 | 1956
    Hispanic or Latino | 49 | 49 | 98
    Not Hispanic or Latino | 921 | 937 | 1858
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants who had baseline race data.
  Participants
    number analyzed (Participants) | 970 | 986 | 1956
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 75 | 71 | 146
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 14 | 19 | 33
    White | 878 | 894 | 1772
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 61 | 66 | 127
  Sweden | 26 | 26 | 52
  United States | 537 | 541 | 1078
  Japan | 67 | 65 | 132
  Poland | 52 | 50 | 102
  Italy | 46 | 52 | 98
  United Kingdom | 45 | 44 | 89
  Australia | 32 | 36 | 68
  France | 87 | 86 | 173
  Germany | 48 | 48 | 96
  Spain | 56 | 58 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive 14 Item Subscore (ADAS-Cog14)
Description: The ADAS is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS that was used as the primary efficacy measure consists of 14 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation, and maze completion measures. The ADAS-Cog14 scale ranges from 0 to 90. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 1053 | 1067
Units on a scale | 6.65 (0.355) | 7.44 (0.356)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Test type: Superiority; p = 0.095, Mixed Models Analysis; The Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.73 to 0.14]

2. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study- Instrumental Activities of Daily Living (ADCS-iADL)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The total score ranges from 0 to 78, with lower scores indicating greater disease severity. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 908 | 896
Units on a scale | -6.17 (0.318) | -7.17 (0.320)

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive 11 Item Subscore (ADAS-Cog11)
Description: The cognitive subscale of ADAS (ADAS Cog11) consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 1053 | 1067
Units on a scale | 5.22 (0.284) | 5.90 (0.285)

4. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE)
Description: MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 893 | 876
Units on a scale | -3.17 (0.154) | -3.66 (0.156)

5. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL)
Description: as for outcome 2
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 908 | 897
Units on a scale | -7.42 (0.386) | -8.77 (0.387)

6. Secondary Outcome: Change From Baseline in Functional Activities Questionnaire (FAQ)
Description: FAQ is a 10-item, caregiver-based questionnaire and was administered to the study partner who was asked to rate the participant's ability to perform a variety of activities ranging from financial management, shopping, playing games, food preparation, traveling, keeping appointments, keeping track of current events, and understanding media. FAQ total score was calculated by adding the scores from each of the 10 items. A negative change indicated an improvement from baseline. FAQ Total Score is the sum of 10 items, ranging from 0 (best possible outcome) to 100 (worst possible outcome). LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 907 | 892
Units on a scale | 5.17 (0.212) | 5.57 (0.213)

7. Secondary Outcome: Change From Baseline in Clinical Dementia Rating-Sum of Boxes (CDR-SB)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 903 | 895
Units on a scale | 1.91 (2.442) | 2.23 (2.692)

8. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI)
Description: NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the participant's behavior. Total score ranges from 12 to 144; Higher scores indicate greater disease severity. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 909 | 891
Units on a scale | 2.26 (3.11) | 0.382 (0.387)

9. Secondary Outcome: Change From Baseline in Resource Utilization in Dementia-Lite (RUD-Lite)
Description: Assesses healthcare resource utilization (formal and informal care). Information gathered on both caregivers (care-giving time, work status) and participants (accommodation and healthcare resource utilization) was gathered from baseline and follow-up interviews. Reported number of hospitalizations per participant up to 76 weeks. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Number of hospitalizations
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 909 | 891
Number of hospitalizations
  Basic ADL | 0.34 (0.058) | 0.35 (0.058)
  Instrumental ADL | 0.55 (0.099) | 0.50 (0.100)
  Sum of Basic and Instrumental ADL | 0.91 (0.132) | 0.86 (0.134)
  Supervision | 0.72 (0.125) | 0.88 (0.127)

10. Secondary Outcome: Change From Baseline in Quality of Life in Alzheimer's Disease (QoL-AD)
Description: Assesses QoL for AD: participant rates mood, relationships, memory, finances, physical condition, and overall QoL assessment. Each of 13 items, rated on a 4-point scale. Sum of items=total score (range: 13 to 52). Higher scores indicate greater QoL. Participant's primary caregiver asked to complete same measure. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 853 | 812
Units on a scale | -0.55 (0.158) | -0.72 (0.161)

11. Secondary Outcome: Change From Baseline in 5-Dimensional EuroQol Quality of Life Scale Proxy Version (EQ-5D Proxy)
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 3 severity levels: no, some, severe problems. Visual analog scale (VAS) assesses caregiver's impression of participant's health state; score ranges: 0 to 100 millimeter (mm). Lower scores=greater disease severity LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 904 | 892
mm | -1.10 (0.556) | -2.61 (0.562)

12. Secondary Outcome: Change From Baseline in Integrated Alzheimer's Disease Rating Scale (iADRS)
Description: Integrated Alzheimer's Disease Rating Scale is used to assess that solanezumab slows down the cognitive and functional decline associated with AD compared with placebo. iADRS is a simple linear combination of ADAS-Cog 13 or 14 and the ADCS-iADL. The scale ranges from 0 to 146, where lower scores indicate worse performance. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 903 | 883
units on a scale | -12.92 (0.533) | -14.59 (0.537)

13. Secondary Outcome: Percentage of Participants of Cognitive and Functional Responders
Description: Assess the proportion of participants who reach certain levels of cognitive and functional decline. Decline in cognition was defined as worsening from baseline by at least 6 or 9 points on the ADAS Cog14. If there is a cognitive decline of a specified cut-off or more at any time then the participant is considered a nonresponder. Functional nonresponders are participants who have not had any of the following at any time point: Clinically evident decline in ability to perform one or more basic ADL present at baseline; A clinically evident decline in ability to perform 20% or more of the instrumental ADL present at baseline; An increase in global CDR score of 1 point or more compared with baseline. A decline from no impairment to mild impairment (bADL, iADL is not considered clinically significant, but other declines of 1 or more points and any participant discontinuation within the first 6 months will be considered a non-responder.
Time Frame: Baseline through Week 80
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 1057 | 1072
percentage of participants
  Cognitive Responders: Cut-off 6 | 35.7 | 35.3
  Cognitive Responders: Cut-off 9 | 55.2 | 52.3
  Functional Responders | 38.0 | 36.8

14. Secondary Outcome: Change From Baseline in Plasma Amyloid-Beta (Aβ) Species
Description: Concentration of amino acid peptide known as Aβ 1-42 in plasma. The change in plasma Aβ analytes after treatment were assessed separately for each plasma Aβ parameter. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Picogram/milliliter
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 1057 | 1072
Picogram/milliliter
  Modified amyloid beta 1-40: number analyzed (Participants) | 841 | 842
  Modified amyloid beta 1-40 | 172754.36 (1613.534) | 262.98 (1609.006)
  Modified amyloid beta1-42: number analyzed (Participants) | 848 | 840
  Modified amyloid beta1-42 | 18485.26 (104.913) | 15.75 (105.237)

15. Secondary Outcome: Change From Baseline in Volumetric Magnetic Resonance Imaging (vMRI)
Description: The vMRI assessment of right and left hippocampal atrophy, is reported. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Cubic millimeter (mm^3)
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 1057 | 1072
Cubic millimeter (mm^3)
  Right hippocampal atrophy: number analyzed (Participants) | 789 | 771
  Right hippocampal atrophy | -145.7 (75.42) | -154.1 (81.06)
  Left hippocampal atrophy: number analyzed (Participants) | 789 | 771
  Left hippocampal atrophy | -142.3 (74.27) | -146.3 (78.04)
  Right hippocampal atrophy+Left hippocampal atrophy: number analyzed (Participants) | 789 | 771
  Right hippocampal atrophy+Left hippocampal atrophy | -288.0 (135.19) | -300.4 (138.52)
  Right entorhinal cortex atrophy: number analyzed (Participants) | 789 | 771
  Right entorhinal cortex atrophy | -77.3 (45.18) | -80.8 (45.16)
  Left entorhinal cortex atrophy: number analyzed (Participants) | 789 | 771
  Left entorhinal cortex atrophy | -91.6 (47.60) | -95.2 (53.46)
  Right+Left entorhinal cortex atrophy: number analyzed (Participants) | 789 | 771
  Right+Left entorhinal cortex atrophy | -169.0 (79.65) | -176.0 (86.11)
  Atrophy of whole brain volume: number analyzed (Participants) | 786 | 769
  Atrophy of whole brain volume | -22725.6 (11920.78) | -23500.5 (12000.09)
  Enlargement of Ventricular volume: number analyzed (Participants) | 788 | 770
  Enlargement of Ventricular volume | 7055.4 (4580.36) | 7226.6 (4545.73)

16. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Solanezumab (LY2062430)
Description: Area Under the Concentration versus Time Curve was evaluated for Solanezumab.
Time Frame: Visit 2 (Post-dose), Visit 5, 9, 15 (Pre-dose, Post-dose) and Visit 22 (Pre-dose): Pre-dose before the infusion, Post-dose 30 minutes End of Infusion
Population: All randomized participants who received at least 1 dose of study medication (Solanezumab) with evaluable Solanezumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram*hour per milliliter (mg*h/mL)
Arm/Group | Solanezumab
Number analyzed (Participants) | 1044
milligram*hour per milliliter (mg*h/mL) | 43.2 (24.3)

17. Secondary Outcome: Change From Baseline in Florbetapir Positron Emission Tomography (PET) Scan
Description: Florbetapir PET imaging was used to confirm the presence of amyloid pathology consistent with AD. Change from baseline was done to test the hypothesis that amyloid burden was reduced in participants in the treatment group. The change from baseline to the postbaseline visit of the composite summary standard uptake value ratio of florbetapir F18 was calculated. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit. The composite summary measure is an unweighted average of the 6 smaller regions (anterior cingulate, frontal medial orbital, parietal, posterior cingulate, precuneus, and temporal) normalized to whole cerebellum or subject-specific white matter.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: standard uptake value ratio
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 915 | 924
standard uptake value ratio
  Subject specific white matter corrected: number analyzed (Participants) | 805 | 791
  Subject specific white matter corrected | 0.02 (0.002) | 0.02 (0.002)
  Mean whole cerebellum corrected: number analyzed (Participants) | 805 | 791
  Mean whole cerebellum corrected | -0.01 (0.005) | 0.00 (0.005)

18. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Aβ Levels
Description: Concentration of CSF parameters includes amino acid peptide known as Aβ 1-42 and Aβ 1-42. Analyses of these CSF biomarkers was conducted in a subset of participants (as an addendum to the protocol). The dependent variable for each CSF parameter was its change from baseline to endpoint. LS Mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit.
Time Frame: Baseline, Week 80
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline data.
Measure: Least Squares Mean (Standard Error); unit: picogram/milliliter
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 1057 | 1072
picogram/milliliter
  Free amyloid beta 1-42, CSF | -37.33 (7.507) | -9.27 (8.175)
  Modified amyloid beta 1-42, CSF | 315.69 (42.620) | -107.91 (42.907)

ADVERSE EVENTS:
Time Frame: Up To 80 Weeks
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- Solanezumab: Double-Blind Phase: Participants received Solanezumab 400 mg IV every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who completed the full 80 weeks of treatment/assessment and decide to continue will take this regimen for up to an additional 208 weeks.
- Placebo: Double-Blind Phase: Participants received Placebo IV every 4 weeks for 76 weeks with an additional 4 weeks of assessments. Participants who complete the full 80 weeks of treatment/assessment and decide to continue will switch to solanezumab 400 mg every 4 weeks for up to an additional 208 weeks.
- Solanezumab: Open Label: Participants who complete 80 weeks treatment/assessment of the double-blind period were entered into open-label period. Participants received Solanezumab 400 mg IV every 4 weeks for 180 weeks with an additional 4 weeks of assessments.
- Placebo: Open Label: Participants who complete 80 weeks treatment/assessment of the double-blind period were entered into open-label period. Participants received Placebo IV every 4 weeks for 180 weeks with an additional 4 weeks of assessments.
Arm/Group | Solanezumab: Double-Blind Phase | Placebo: Double-Blind Phase | Solanezumab: Open Label | Placebo: Open Label
Serious Adverse Events (participants affected / at risk) | 175/1054 | 203/1067 | 102/879 | 114/856
Other Adverse Events (participants affected / at risk) | 536/1054 | 530/1067 | 255/879 | 260/856
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Solanezumab: Double-Blind Phase (N=1054) | Placebo: Double-Blind Phase (N=1067) | Solanezumab: Open Label (N=879) | Placebo: Open Label (N=856)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Adams-stokes syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 9 (9) | 4 (4) | 5 (5)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 7 (8) | 5 (7) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical mycobacterial pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0/455 (0) | 0/440 (0) | 0/378 (0) | 1/348 (1)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraspinal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 11 (11) | 8 (8) | 3 (3) | 5 (5)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 8 (9) | 2 (2) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 24 (26) | 24 (27) | 5 (5) | 12 (12)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 6 (7) | 5 (5) | 3 (3) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6) | 3 (3) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin t increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 3 (3) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/599 (0) | 1/627 (1) | 0/501 (0) | 0/508 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/599 (0) | 1/627 (1) | 0/501 (0) | 0/508 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/455 (2) | 0/440 (0) | 2/378 (2) | 0/348 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/455 (1) | 1/440 (1) | 0/378 (0) | 1/348 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell cancer of renal pelvis and ureter metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/599 (1) | 0/627 (0) | 0/501 (0) | 0/508 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 5 (7) | 0 (0) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dementia alzheimer's type (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Dementia of the alzheimer's type, with delirium (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 8 (11) | 14 (14) | 5 (5) | 7 (7)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (3)
Phobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/455 (1) | 1/440 (1) | 3/378 (3) | 0/348 (0)
Prostatitis (Reproductive system and breast disorders) | 1/455 (1) | 0/440 (0) | 0/378 (0) | 0/348 (0)
Vulvar dysplasia (Reproductive system and breast disorders) | 0/599 (0) | 1/627 (1) | 0/501 (0) | 0/508 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immobilisation prolonged (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respite care (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solanezumab: Double-Blind Phase (N=1054) | Placebo: Double-Blind Phase (N=1067) | Solanezumab: Open Label (N=879) | Placebo: Open Label (N=856)
Diarrhoea (Gastrointestinal disorders) | 76 (86) | 87 (109) | 23 (24) | 17 (18)
Nausea (Gastrointestinal disorders) | 54 (69) | 46 (63) | 23 (32) | 15 (18)
Nasopharyngitis (Infections and infestations) | 89 (114) | 80 (99) | 29 (31) | 32 (36)
Upper respiratory tract infection (Infections and infestations) | 64 (74) | 54 (61) | 23 (25) | 21 (23)
Urinary tract infection (Infections and infestations) | 58 (79) | 72 (103) | 38 (47) | 36 (46)
Fall (Injury, poisoning and procedural complications) | 146 (195) | 144 (207) | 67 (97) | 80 (109)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (51) | 56 (62) | 21 (23) | 22 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 63 (70) | 60 (67) | 26 (26) | 23 (23)
Dizziness (Nervous system disorders) | 61 (66) | 57 (65) | 23 (24) | 29 (31)
Headache (Nervous system disorders) | 86 (96) | 86 (151) | 28 (34) | 29 (42)
Anxiety (Psychiatric disorders) | 54 (57) | 58 (59) | 15 (18) | 17 (17)
Depression (Psychiatric disorders) | 60 (62) | 57 (57) | 18 (18) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (53) | 58 (69) | 25 (27) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.